CLINICAL TRIAL: NCT00727779
Title: Mechanisms by Which Strength Training Ameliorates the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Charles A. Stuart, Professor, Internal Medicine, East Tennessee State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R15DK080488 (NIH); R15DK080488 (NIH)
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Metabolic Syndrome
Keywords: diabetes, metabolic syndrome, type 2 diabetes
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metabolic syndrome (Experimental): intervention is to undergo eight weeks of progressive strength training; metabolic syndrome subjects will have baseline and post-intervention assessments including muscle biopsies and insulin clamps
  Interventions: Behavioral: strength training
- control subjects (Active Comparator): intervention is to undergo eight weeks of progressive strength training; non-obese sedentary subjects will have the same assessments as the metabolic syndrome subjects and exercise training simultaneously.
  Interventions: Behavioral: strength training

INTERVENTIONS:
Behavioral: strength training — eight weeks of progressively increasing resistance training will be done in both groups side-by-side

SUMMARY:
Prevention and treatment strategies for diabetes use exercise as the cornerstone. Even though endurance training and strength training both improve insulin resistance, strength training may be better suited for persons at risk for type 2 diabetes. We will expand our pilot studies of muscle adaptation induced by resistance exercise training to determine the biochemical mechanisms that will cause people with the Metabolic Syndrome to secure major benefit from intense strength training.

DETAILED DESCRIPTION:
Life style alterations can be powerful deterrents to developing type 2 diabetes and are cornerstones of the treatment of this condition. Both aerobic and resistance exercise improve diabetes blood glucose control and insulin resistance. These two types of exercise appear to exert their effects on different muscle fiber types - red for endurance and white for strength. Similar to the effects of endurance exercise training, strength training increases muscle glucose transporter isoform 4 (GLUT4), but in contrast, mitochondria numbers do not increase. We hypothesize (1) that strength training in persons with pre-diabetes may be effective in reversing insulin resistance by novel mechanisms that are distinct from the endurance training-induced mitochondrial biogenesis. We further hypothesize (2) that resistance exercise training enhances whole body insulin action primarily by increasing the white fiber size via the protein kinase mammalian target of rapamycin (mTOR) and improves insulin-stimulated glucose uptake by increased GLUT4 expression primarily in white fibers of the trained muscles. In this proposal, we will perform eight weeks of progressive strength training on ten subjects with the Metabolic Syndrome who are at high risk for developing type 2 diabetes and on ten sedentary control subjects. This project builds on our experience with a study of focused resistance training whose results are presented in this application. In this pilot study, subjects exercised on stationary bicycles for six weeks causing muscle GLUT4 and phopho-mTOR to increase substantially, but maximal oxygen uptake (VO2max), phospho-AMP-activated protein kinase (AMPK), peroxisome proliferator-activated receptor-γ co-activator (PGC-1α), and mitochondrial markers did not change. Our hypotheses will be tested by two Specific Aims. (1) Subjects at high risk for diabetes will undergo progressively increasing intensity resistance exercise training and increased strength and improved insulin responsiveness will both be quantified to demonstrate significant benefit, and (2) quantify the effect of resistance exercise training on anatomic and functional adaptation in muscle. We will characterize fiber type, fiber size, fiber-specific changes in mitochondrial DNA and enzymes, fiber-specific changes in the principle glucose transporters in muscle (GLUT4, GLUT5, and GLUT12), and evaluate changes in two distinct intramuscular pathways (AMPK, mTOR) and regulatory factors (PGC-1α, PPARγ, PPARδ) using immunoblots of muscle subcellular fractions and immunohistochemical techniques. These evaluations of molecular mechanisms will also include assessing changes in full human Affymetrix gene array data that may move us to new potential resistance training-regulated gene targets. It is the long-term goal of this team of investigators to understand the interplay between life style changes and pharmacological agents in the prevention and treatment of diabetes. Our results will facilitate the development of more effective clinical options to turn back the epidemic of obesity and diabetes in the United States.

ELIGIBILITY:
Inclusion Criteria:

obese family history of diabetes

Exclusion Criteria:

non-obese diabetes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
euglycemic clamp steady state glucose infusion rate (clamp GIR) | pre- post- intervention

SECONDARY OUTCOMES:
GLUT4 content of muscle | pre- post- intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Stuart, MD, Principal Investigator — East Tennessee State University, Johnson City, TN
Locations (1):
- East Tennessee State Univ, Johnson City, Tennessee, United States

REFERENCES:
- [Background] Stuart CA, Yin D, Howell ME, Dykes RJ, Laffan JJ, Ferrando AA. Hexose transporter mRNAs for GLUT4, GLUT5, and GLUT12 predominate in human muscle. Am J Physiol Endocrinol Metab. 2006 Nov;291(5):E1067-73. doi: 10.1152/ajpendo.00250.2006. Epub 2006 Jun 27. PMID 16803853
- [Background] Reeds DN, Stuart CA, Perez O, Klein S. Adipose tissue, hepatic, and skeletal muscle insulin sensitivity in extremely obese subjects with acanthosis nigricans. Metabolism. 2006 Dec;55(12):1658-63. doi: 10.1016/j.metabol.2006.08.006. PMID 17142140
- [Background] Stuart CA, Howell ME, Yin D. Overexpression of GLUT5 in diabetic muscle is reversed by pioglitazone. Diabetes Care. 2007 Apr;30(4):925-31. doi: 10.2337/dc06-1788. Epub 2007 Jan 24. PMID 17251278
- [Background] Moorman J, Zhang Y, Liu B, LeSage G, Chen Y, Stuart C, Prayther D, Yin D. HIV-1 gp120 primes lymphocytes for opioid-induced, beta-arrestin 2-dependent apoptosis. Biochim Biophys Acta. 2009 Aug;1793(8):1366-71. doi: 10.1016/j.bbamcr.2009.05.007. Epub 2009 May 27. PMID 19477204
- [Result] Copland JA, Pardini AW, Wood TG, Yin D, Green A, Bodenburg YH, Urban RJ, Stuart CA. IGF-1 controls GLUT3 expression in muscle via the transcriptional factor Sp1. Biochim Biophys Acta. 2007 Nov-Dec;1769(11-12):631-40. doi: 10.1016/j.bbaexp.2007.08.002. Epub 2007 Sep 4. PMID 17920708
- [Result] Layne AS, Nasrallah S, South MA, Howell ME, McCurry MP, Ramsey MW, Stone MH, Stuart CA. Impaired muscle AMPK activation in the metabolic syndrome may attenuate improved insulin action after exercise training. J Clin Endocrinol Metab. 2011 Jun;96(6):1815-26. doi: 10.1210/jc.2010-2532. Epub 2011 Apr 20. PMID 21508135
- [Result] Stuart CA, Ross IR, Howell ME, McCurry MP, Wood TG, Ceci JD, Kennel SJ, Wall J. Brain glucose transporter (Glut3) haploinsufficiency does not impair mouse brain glucose uptake. Brain Res. 2011 Apr 12;1384:15-22. doi: 10.1016/j.brainres.2011.02.014. PMID 21316350
- [Result] Stuart CA, Howell ME, Cartwright BM, McCurry MP, Lee ML, Ramsey MW, Stone MH. Insulin resistance and muscle insulin receptor substrate-1 serine hyperphosphorylation. Physiol Rep. 2014 Dec 3;2(12):e12236. doi: 10.14814/phy2.12236. Print 2014 Dec 1. PMID 25472611
- [Result] Stuart CA, South MA, Lee ML, McCurry MP, Howell ME, Ramsey MW, Stone MH. Insulin responsiveness in metabolic syndrome after eight weeks of cycle training. Med Sci Sports Exerc. 2013 Nov;45(11):2021-9. doi: 10.1249/MSS.0b013e31829a6ce8. PMID 23669880
- [Result] Stuart CA, McCurry MP, Marino A, South MA, Howell ME, Layne AS, Ramsey MW, Stone MH. Slow-twitch fiber proportion in skeletal muscle correlates with insulin responsiveness. J Clin Endocrinol Metab. 2013 May;98(5):2027-36. doi: 10.1210/jc.2012-3876. Epub 2013 Mar 20. PMID 23515448